CLINICAL TRIAL: NCT02096263
Title: Immunogenicity and Safety Study of GSK Biologicals' Infanrix Hexa at 2, 4 and 6 Months of Age in Healthy Infants
Brief Title: Study to Determine the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals; Infanrix Hexa at 2, 4 and 6 Months of Age in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 117119; 2013-004304-19 (EudraCT Number)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Poliomyelitis; Diphtheria; Haemophilus Influenzae Type b; Tetanus; Acellular Pertussis; Hepatitis B
Keywords: Infants; Safety; Healthy; Infanrix Hexa; Immunogenicity
MeSH Terms: conditions — Poliomyelitis; Diphtheria; Haemophilus Infections; Tetanus; Hepatitis B | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; PEDIARIX; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; pentacel; Engerix-B; Diphtheria-Tetanus-acellular Pertussis Vaccines; Hiberix; RIX4414 vaccine

ARMS (3):
- Infanrix hexa Group (Experimental): Subjects between, and including, 6 and 12 weeks of age at the time of the vaccination received, in the Primary Phase of the study, 3 doses of Infanrix hexa (lot A, lot B or lot C as per the group allocation) co-administered with Prevnar13 at 2, 4 and 6 months of age and Rotarix at 2 and 4 months of age. The injectable vaccines were administered by intramuscular injection in the anterolateral thigh, while Rotarix was administered orally. Subjects received a booster dose of Infanrix and Hiberix at 15-18 months of age by intramuscular injection in the anterolateral thigh.
  Interventions: Biological: Infanrix hexa; Biological: Infanrix; Biological: Hiberix; Biological: Prevnar13; Biological: Rotarix
- Pediarix Group (Active Comparator): Subjects between, and including, 6 and 12 weeks of age at the time of the vaccination received, in the Primary Phase of the study, 3 doses of Pediarix and ActHIB co-administered with Prevnar13 at 2, 4 and 6 months of age and Rotarix at 2 and 4 months of age. The injectable vaccines were administered by intramuscular injection in the anterolateral thigh, while Rotarix was administered orally. Subjects received a booster dose of Infanrix and ActHIB at 15-18 months of age by intramuscular injection in the anterolateral thigh.
  Interventions: Biological: Pediarix; Biological: ActHIB; Biological: Infanrix; Biological: Prevnar13; Biological: Rotarix
- Pentacel Group (Active Comparator): Subjects between, and including, 6 and 12 weeks of age at the time of the vaccination received, in the Primary Phase of the study, 3 doses of Pentacel and Engerix co-administered with Prevnar13 at 2, 4 and 6 months of age and Rotarix at 2 and 4 months of age. The injectable vaccines were administered by intramuscular injection in the anterolateral thigh, while Rotarix was administered orally. Subjects received a booster dose of Pentacel at 15-18 months of age by intramuscular injection in the anterolateral thigh.
  Interventions: Biological: Pentacel; Biological: Engerix-B; Biological: Prevnar13; Biological: Rotarix

INTERVENTIONS:
Biological: Infanrix hexa — 3 doses administered intramuscularly in the right thigh.
  Arms: Infanrix hexa Group
Biological: Pediarix — 3 doses administered intramuscularly in the right thigh
  Arms: Pediarix Group
Biological: ActHIB — 4 doses administered intramuscularly in the upper left thigh
  Arms: Pediarix Group
Biological: Pentacel — 4 doses administered intramuscularly in the right thigh
  Arms: Pentacel Group
Biological: Engerix-B — 2 or 3 doses administered intramuscularly in the upper left thigh
  Arms: Pentacel Group
Biological: Infanrix — 1 dose administered intramuscularly in the right thigh
  Arms: Infanrix hexa Group; Pediarix Group
Biological: Hiberix — 1 dose administered intramuscularly in the left thigh
  Arms: Infanrix hexa Group
Biological: Prevnar13 — 3 doses administered intramuscularly in the lower left thigh
Biological: Rotarix — 2 doses administered orally

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of GSK Biologicals' Infanrix hexa vaccine when administered to healthy infants as primary vaccination at 2, 4 and 6 months of age, co-administered with Prevnar and Rotarix with a booster dose of GSK Biologicals' Infanrix and Hiberix vaccines at 15-18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/ Legally Acceptable Representative(s) (LARs) who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Born full-term (i.e. after a gestation period of 37 weeks to less than 42 completed weeks [259 to 293 days]).
* Written informed consent obtained from parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Infants who have not received a previous dose of hepatitis B vaccine or those who have received only 1 dose of hepatitis B vaccine administered at least 30 days prior to enrolment.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccines, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting from 30 days before the first vaccination until 30 days after Dose 3 (Epoch 001, primary vaccination) and from 30 days before the booster Dose 4 until 30 days after booster Dose 4 (Epoch 002, booster vaccination), i.e. the end of the study:

  * Inactivated influenza and hepatitis A vaccines are allowed throughout the study.
  * Routine administration(s) of vaccines are allowed from 30 days after the last dose of primary vaccination until 30 days before the booster dose and after post-booster blood sampling. Routine administration of measles-mumps-rubella vaccine, varicella, pneumococcal vaccines are allowed from 30 days after last dose of primary vaccine until 30 days before booster dose and from post-booster blood sampling, as well as according to the recommended immunization schedule in US.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* History of Hib, diphtheria, tetanus, pertussis, pneumococcal, rotavirus, poliovirus and hepatitis B diseases.
* Previous vaccination against Hib, diphtheria, tetanus, pertussis, pneumococcus, rotavirus and/or poliovirus; more than one previous dose of hepatitis B vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines (including yeast).
* Hypersensitivity to latex.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders including seizures.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* History of intussusception or of any uncorrected congenital malformation of the gastrointestinal tract that would predispose the infant to intussusception.
* History of Severe Combined Immunodeficiency Disease (SCID).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥38.0°C /100.4°F by any route. The preferred route for recording temperature in this study will be rectal for Epoch 001 and axillary for Epoch 002.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 585 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2015-02-06 (Actual); Study Completion 2015-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (41):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Orange City, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Augusta, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Nicholasville, Kentucky
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Payson, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Ellensburg, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=19670

REFERENCES:
- [Background] Klein NP, Abu-Elyazeed R, Cheuvart B, Janssens W, Mesaros N. Immunogenicity and safety following primary and booster vaccination with a hexavalent diphtheria, tetanus, acellular pertussis, hepatitis B, inactivated poliovirus and Haemophilus influenzae type b vaccine: a randomized trial in the United States. Hum Vaccin Immunother. 2019;15(4):809-821. doi: 10.1080/21645515.2018.1549449. Epub 2019 Jan 4. PMID 30444673
- See also: Full CSR redacted with additional report posting on GSK. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=117119&attachmentIdentifier=f37b4392-6468-49a6-9f43-ebda8ddbc0f1&fileName=gsk-117119-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 43 centers in the United States of America (USA).
Period: Overall Study
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Started | 195 | 194 | 196
Completed | 161 | 158 | 157
Not Completed | 34 | 36 | 39
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 14 | 18 | 15
Not completed — Other | 7 | 9 | 6
Not completed — Sponsor study termination | 0 | 0 | 1
Not completed — Protocol Violation | 7 | 2 | 8
Not completed — Withdrawal by Subject | 5 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group | Total
Number analyzed (Participants) | 195 | 194 | 196 | 585
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.5 (1.0) | 8.6 (1.1) | 8.6 (1.1) | 8.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 80 | 95 | 276
  Male | 94 | 114 | 101 | 309
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese Heritage | 1 | 0 | 1 | 2
  African Heritage / African American | 16 | 9 | 20 | 45
  Asian - East Asian Heritage | 3 | 2 | 0 | 5
  White - Caucasian / European Heritage | 118 | 128 | 115 | 361
  Asian - Central/South Asian Heritage | 2 | 2 | 1 | 5
  White - Arabic / North African Heritage | 0 | 1 | 0 | 1
  Unspecified | 29 | 27 | 32 | 88
  American Indian or Alaskan Native | 15 | 15 | 17 | 47
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 2 | 5
  Asian - South East Asian Heritage | 9 | 9 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations for Pertussis Toxoid (Anti-PT), Filamentous Hemagglutinin (Anti-FHA) and Pertactin (Anti-PRN).
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the following cut-offs:2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA, and 2.187 IU/mL for anti-PRN. The results for the Infanrix hexa Group and Pediarix Group were the primary outcome variables.
Time Frame: At Month 5, one month after the third dose of the primary vaccination.
Population: The analysis was done on the Primary According to Protocol (ATP) cohort for immunogenicity, which included all subjects who complied with the protocol up to the post-dose 3 blood sample and who had immunogenicity results for the post-dose 3 blood sample.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 146 | 149 | 149
IU/mL
  Anti-PT | 43.2 [38.1 to 48.9] | 48.3 [42.7 to 54.5] | 24.2 [21.1 to 27.7]
  Anti-FHA | 106.3 [95.0 to 119.0] | 122.7 [109.9 to 137.0] | 59.9 [51.7 to 69.3]
  Anti-PRN | 57.4 [49.5 to 66.6] | 46.9 [39.9 to 55.3] | 33.0 [27.8 to 39.1]
Statistical Analysis 1: Comparison: Infanrix Hexa Group vs Pediarix Group; To demonstrate the non-inferiority of Infanrix hexa to Pediarix co-administered with ActHIB, in terms of antibody geometric mean concentrations (GMCs) for pertussis antigen, pertussis toxoid (PT), one month after the third dose of the primary vaccination; Test type: Non-Inferiority — Non-inferiority in terms of immune response to pertussis antigens will be demonstrated if, for each of the three antigens, the upper limit of the 95% confidence interval (CI) on the GMC ratio [Pediarix Group divided by Infanrix hexa Group] is ≤ 1.5; Adjusted GMC ratio = 1.1, 95% CI 2-sided [0.92 to 1.31] — Adjusted GMC (ANCOVA model adjusted with the vaccine group as fixed effect and the Infanrix vaccination history of the mother during pregnancy as continuous regressor)
Statistical Analysis 2: Comparison: Infanrix Hexa Group vs Pediarix Group; To demonstrate the non-inferiority of Infanrix hexa to Pediarix co-administered with ActHIB, in terms of antibody geometric mean concentrations (GMCs) for pertussis antigen, filamentous hemagglutinin (FHA), one month after the third dose of the primary vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 1.14, 95% CI 2-sided [0.97 to 1.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Infanrix Hexa Group vs Pediarix Group; To demonstrate the non-inferiority of Infanrix hexa to Pediarix co-administered with ActHIB, in terms of antibody geometric mean concentrations (GMCs) for pertussis antigen, pertactin (PRN), one month after the third dose of the primary vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.79, 95% CI 2-sided [0.63 to 0.99] — Adjusted GMC (ANCOVA model adjusted with the vaccine group as fixed effect and the Tdap vaccination history of the mother during pregnancy as continuous regressor.)

2. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN.
Description: A seropositive subject was defined as a subject with antibody concentrations above to or equal to (≥) 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA, and 2.187 IU/mL for anti-PRN.
Time Frame: At Month 5, one month after the third dose of the primary vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 146 | 149 | 149
Participants
  Anti-PT | 146 | 148 | 148
  Anti-FHA | 146 | 149 | 149
  Anti-PRN | 146 | 148 | 148

3. Secondary Outcome: Number of Seroprotected Subjects Against Tetanus (T).
Description: A seroprotected subject was defined a a subject with antibody concentrations ≥ 0.1 IU/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 146 | 149 | 149
Participants | 146 | 149 | 148

4. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (D).
Description: A seroprotected subject was defined a a subject with antibody concentrations ≥ 0.1 IU/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 142 | 144 | 149
Participants | 142 | 144 | 149

5. Secondary Outcome: Antibody Concentrations for Anti-T.
Description: Concentrations were expressed as GMCs for the seroprotection cut-off of 0.1 IU/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 146 | 149 | 149
IU/mL | 2.458 [2.195 to 2.753] | 2.633 [2.338 to 2.966] | 2.012 [1.768 to 2.290]

6. Secondary Outcome: Antibody Concentrations for Anti-D.
Description: Concentrations were expressed as GMCs for the seroprotection cut-off of 0.1 IU/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 142 | 144 | 149
IU/mL | 1.777 [1.551 to 2.036] | 1.648 [1.44 to 1.886] | 1.249 [1.095 to 1.425]

7. Secondary Outcome: Number of Seroprotected Subjects Against Anti-polio Types 1, 2 and 3.
Description: A seroprotected subject was defined as a subject with anti-polio types 1, 2 and 3 titres ≥ 8 dilution.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 137 | 134 | 136
Participants
  Anti-polio 1 | 137 | 134 | 135
  Anti-polio 2: number analyzed (Participants) | 133 | 131 | 134
  Anti-polio 2 | 133 | 131 | 134
  Anti-polio 3: number analyzed (Participants) | 129 | 132 | 126
  Anti-polio 3 | 129 | 132 | 124

8. Secondary Outcome: Antibody Titres for Anti-polio Types 1, 2 and 3.
Description: Titres were expressed as geometric mean titres (GMTs) for the cut-off of 8 dilution.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titres
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 137 | 134 | 136
titres
  Anti-polio 1 | 546.9 [447.7 to 668.0] | 604.1 [495.9 to 736.0] | 319.5 [256.8 to 397.5]
  Anti-polio 2: number analyzed (Participants) | 133 | 131 | 134
  Anti-polio 2 | 483.5 [394.2 to 593.0] | 567.7 [448.8 to 718.1] | 283.0 [229.4 to 349.2]
  Anti-polio 3: number analyzed (Participants) | 129 | 132 | 126
  Anti-polio 3 | 722.2 [577.4 to 903.4] | 927.0 [740.7 to 1160.3] | 294.6 [221.6 to 391.7]

9. Secondary Outcome: Number of Seroprotected Subjects Against Polyribosyl Ribitol Phosphate (Anti-PRP).
Description: A seroprotected subject was defined as a subject with anti-PRP concentrations ≥ 0.15 µg/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 154 | 154 | 156
Participants | 146 | 151 | 154

10. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 1 µg/mL.
Description: The cut-off for this assay was an anti-PRP concentration ≥ 1 µg/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 154 | 154 | 156
Participants | 85 | 145 | 130

11. Secondary Outcome: Antibody Concentrations for Anti-PRP.
Description: Antibody concentrations were expressed as GMCs for the assay cut-off of 1 µg/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 154 | 154 | 156
µg/mL | 1.348 [1.076 to 1.688] | 9.258 [7.362 to 11.642] | 5.717 [4.363 to 7.492]

12. Secondary Outcome: Number of Seroprotected Subjects Against Hepatitis B (Anti-HBs).
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mili-International units per mililiter (mIU/mL).
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 134 | 138 | 136
Participants | 134 | 138 | 133

13. Secondary Outcome: Antibody Concentrations for Anti-HBs.
Description: Antibody concentrations were expressed as GMCs for the seroprotection cut-off of 10 mIU/mL.
Time Frame: At Month 5, one month after the third dose of the primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 134 | 138 | 136
mIU/mL | 2258.8 [1910.7 to 2670.4] | 1886.0 [1565.6 to 2271.9] | 1053.4 [780.2 to 1422.4]

14. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: The solicited local symptoms assessed were pain, redness and swelling. Any = any reports of the specific symptom irrespective of intensity grade; above or equal (≥); Grade 2 Redness/Swelling: > 5 millimeters (mm); Grade 3 Redness/Swelling: > 20 mm; Grade 2 Pain = Moderate: cries/protests on touch; Grade 3 Pain = Severe: Cries when limb is moved/spontaneously painful. Grade = G; Medical Advice = MA.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following Dose 1
Population: The analysis was done on the Primary Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and who had their symptoms sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 185 | 189 | 188
Participants
  Any Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 123 | 100
  ≥ G 2 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 66 | 45
  G 3 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 22 | 10
  MA Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  Any Pain, Infanrix hexa/Pediarix/Pentacel | 94 | 113 | 115
  ≥ G 2 Pain, Infanrix hexa/Pediarix/Pentacel | 40 | 65 | 51
  G 3 Pain, Infanrix hexa/Pediarix/Pentacel | 8 | 17 | 12
  MA Pain, Infanrix hexa/Pediarix/Pentacel | 1 | 0 | 0
  Any Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 63 | 55
  ≥ G 2 Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 19 | 12
  G 3 Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 8 | 1
  MA Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  Any Redness, Infanrix hexa/Pediarix/Pentacel | 47 | 56 | 57
  ≥ G 2 Redness, Infanrix hexa/Pediarix/Pentacel | 15 | 15 | 20
  G 3 Redness, Infanrix hexa/Pediarix/Pentacel | 3 | 4 | 3
  MA Redness, Infanrix hexa/Pediarix/Pentacel | 0 | 0 | 0
  Any Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 41 | 39
  ≥ G 2 Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 14 | 14
  G 3 Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 6 | 3
  MA Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  Any Swelling, Infanrix hexa/Pediarix/Pentacel | 31 | 35 | 45
  ≥ G 2 Swelling, Infanrix hexa/Pediarix/Pentacel | 10 | 14 | 24
  G 3 Swelling, Infanrix hexa/Pediarix/Pentacel | 2 | 3 | 11
  MA Swelling, Infanrix hexa/Pediarix/Pentacel | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: The solicited local symptoms assessed were pain, redness (Red) and swelling (Swe). Any = any reports of the specific symptom irrespective of intensity grade; above or equal (≥); Grade 2 Redness/Swelling: > 5 millimeters (mm); Grade 3 Redness/Swelling: > 20 mm; Grade 2 Pain = Moderate: cries/protests on touch; Grade 3 Pain = Severe: Cries when limb is moved/spontaneously painful. Grade = G; Medical Advice = MA.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following Dose 2
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 182 | 184 | 180
Participants
  Any Pain, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  Any Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 104 | 6
  ≥ G 2 Pain, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  ≥ G 2 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 47 | 2
  G 3 Pain, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  G 3 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 9 | 0
  MA Pain, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  MA Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 0 | 0
  Any Pain,Infanrix/Pediarix/Pentacel | 84 | 108 | 93
  ≥G2 Pain,Infanrix/Pediarix/Pentacel | 25 | 44 | 31
  G3 Pain,Infanrix/Pediarix/Pentacel | 1 | 7 | 6
  MA Pain, Infanrix/Pediarix/Pentacel | 0 | 0 | 0
  Any Redness, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  Any Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 66 | 5
  ≥ G 2 Redness, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  ≥ G 2 Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 17 | 1
  G 3 Redness, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  G 3 Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  MA Redness, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  MA Redness, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 0 | 0
  Any Red, Infanrix/Pediarix/Pentacel | 59 | 61 | 64
  ≥G2 Red,Infanrix/Pediarix/Pentacel | 15 | 12 | 15
  G 3 Red, Infanrix/Pediarix/Pentacel | 3 | 3 | 2
  MA Red, Infanrix/Pediarix/Pentacel | 0 | 0 | 0
  Any Swelling, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  Any Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 40 | 3
  ≥ G 2 Swelling, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  ≥ G 2 Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 11 | 0
  G 3 Swelling, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  G 3 Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  MA Swelling, ActHIB/Engerix: number analyzed (Participants) | 182 | 184 | 13
  MA Swelling, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 0 | 0
  Any Swe, Infanrix/Pediarix/Pentacel | 41 | 40 | 42
  ≥G2 Swe, Infanrix/Pediarix/Pentacel | 10 | 12 | 7
  G 3 Swe, Infanrix/Pediarix/Pentacel | 2 | 2 | 3
  MA Swe, Infanrix/Pediarix/Pentacel | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: The solicited local symptoms assessed were pain, redness and swelling. Any = any reports of the specific symptom irrespective of intensity grade; above or equal (≥); Grade 2 Redness/Swelling: > 5 millimeters (mm); Grade 3 Redness (Red)/Swelling (Swe): > 20 mm; Grade 2 Pain = Moderate: cries/protests on touch; Grade 3 Pain = Severe: Cries when limb is moved/spontaneously painful. Grade = G; Medical Advice = MA
Time Frame: During the 4-day (Days 0-3) post-vaccination period following Dose 3
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 172 | 175 | 171
Participants
  Any Pain, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  Any Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 93 | 75
  ≥ G 2 Pain, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  ≥ G 2 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 41 | 25
  G 3 Pain, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  G 3 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 7 | 5
  MA Pain, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  MA Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  Any Pain, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  Any Pain, Infanrix/Pediarix/Pentacel | 67 | 90 | 76
  ≥ G2 Pain, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  ≥ G2 Pain, Infanrix/Pediarix/Pentacel | 18 | 39 | 20
  G3 Pain, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  G3 Pain, Infanrix/Pediarix/Pentacel | 0 | 7 | 7
  MA Pain, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  MA Pain, Infanrix/Pediarix/Pentacel | 0 | 1 | 0
  Any Red, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  Any Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 69 | 51
  ≥ G 2 Red, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  ≥ G 2 Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 7 | 9
  G 3 Red, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  G 3 Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 2
  MA Red, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  MA Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 0 | 0
  Any Red, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  Any Red, Infanrix/Pediarix/Pentacel | 63 | 66 | 56
  ≥G2 Red, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  ≥G2 Red, Infanrix/Pediarix/Pentacel | 7 | 12 | 11
  G3 Red, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  G3 Red, Infanrix/Pediarix/Pentacel | 1 | 3 | 0
  MA Red, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  MA Red, Infanrix/Pediarix/Pentacel | 0 | 1 | 0
  Any Swe, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  Any Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 42 | 37
  ≥ G 2 Swe, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  ≥ G 2 Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 7 | 7
  G 3 Swe, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  G 3 Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  MA Swe, ActHIB/Engerix: number analyzed (Participants) | 172 | 175 | 169
  MA Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 0 | 0
  Any Swe, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  Any Swe, Infanrix/Pediarix/Pentacel | 43 | 44 | 35
  ≥ G2 Swe, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  ≥ G2 Swe, Infanrix/Pediarix/Pentacel | 7 | 10 | 4
  G3 Swe, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  G3 Swe, Infanrix/Pediarix/Pentacel | 1 | 3 | 0
  MA Swe, Infanrix/Pediarix/Pentacel: number analyzed (Participants) | 172 | 175 | 170
  MA Swe, Infanrix/Pediarix/Pentacel | 0 | 1 | 0

17. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: The solicited local symptoms assessed were pain, redness and swelling. Any = any reports of the specific symptom irrespective of intensity grade; above or equal (≥); Grade 2 Redness (Red)/Swelling (Swe): > 5 millimeters (mm); Grade 3 Redness/Swelling: > 20 mm; Grade 2 Pain = Moderate: cries/protests on touch; Grade 3 Pain = Severe: Cries when limb is moved/spontaneously painful. Grade = G; Medical Advice = MA.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following any dose.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 187 | 189 | 188
Participants
  Any Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 148 | 127
  ≥ G 2 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 96 | 62
  G 3 Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 30 | 14
  MA Pain, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 2 | 0
  Any Pain, Infanrix/Pediarix/Pentacel | 127 | 151 | 147
  ≥ G2 Pain, Infanrix/Pediarix/Pentacel | 58 | 93 | 80
  G3 Pain, Infanrix/Pediarix/Pentacel | 8 | 27 | 22
  MA Pain, Infanrix/Pediarix/Pentacel | 1 | 1 | 0
  Any Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 108 | 77
  ≥ G 2 Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 38 | 20
  G 3 Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 10 | 3
  MA Red, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  Any Red, Infanrix/Pediarix/Pentacel | 94 | 98 | 87
  ≥ G2 Red, Infanrix/Pediarix/Pentacel | 27 | 32 | 37
  G3 Red, Infanrix/Pediarix/Pentacel | 7 | 9 | 5
  MA Red, Infanrix/Pediarix/Pentacel | 0 | 1 | 0
  Any Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 78 | 64
  ≥ G 2 Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 25 | 18
  G 3 Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 7 | 3
  MA Swe, ActHIB/Engerix | NA — Subjects in Infanrix hexa Group did not receive the ActHIB or Engerix vaccines. | 1 | 0
  Any Swe, Infanrix/Pediarix/Pentacel | 73 | 70 | 72
  ≥ G2 Swe, Infanrix/Pediarix/Pentacel | 20 | 26 | 26
  G3 Swe, Infanrix/Pediarix/Pentacel | 4 | 7 | 12
  MA Swe, Infanrix/Pediarix/Pentacel | 0 | 1 | 0

18. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: The solicited general symptoms assessed were Drowsiness, Irritability/Fussiness, Loss Of Appetite and Fever (defined as temperature ≥ 38.0°C). Any = any reports of the specific symptom irrespective of intensity grade; Grade 2 (G2) Drowsiness = Drowsiness that interfered with normal activity; Grade 2 Irritability/Fussiness = Moderate: Cried more than usual/interfered with normal activity; Grade 2 Loss of appetite = Ate less than usual/interfered with normal activity; Grade 2 Fever: > 39.0 °C; Grade 3 (G3) Drowsiness/Irritability/Fussiness = symptom that prevented normal activity; Grade 3 Loss of appetite = Did not eat at all; Grade 3 Fever: > 40.0 °C; Related (Rel) = Symptom which was assessed by the investigator as related to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following Dose 1.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 185 | 189 | 188
Participants
  Any Drowsiness | 114 | 143 | 149
  ≥ G 2 Drowsiness | 36 | 56 | 53
  G 3 Drowsiness | 3 | 8 | 12
  Rel Drowsiness | 112 | 136 | 141
  G3 Rel Drowsiness | 3 | 7 | 12
  MA Drowsiness | 1 | 0 | 0
  Any Irritability / Fussiness | 115 | 165 | 153
  ≥ G 2 Irritability / Fussiness | 42 | 79 | 68
  G 3 Irritability / Fussiness | 9 | 17 | 15
  Rel Irritability / Fussiness | 113 | 163 | 147
  G3 Rel Irritability / Fussiness | 9 | 17 | 15
  MA Irritability / Fussiness | 1 | 0 | 0
  Any Loss of appetite | 53 | 76 | 80
  ≥ G 2 Loss of appetite | 8 | 13 | 26
  G 3 Loss of appetite | 0 | 1 | 4
  Rel Loss of appetite | 48 | 73 | 77
  G3 Rel Loss of appetite | 0 | 1 | 4
  MA Loss of appetite | 0 | 0 | 0
  Any Fever | 22 | 34 | 29
  ≥ G 2 Fever | 0 | 0 | 2
  G 3 Fever | 0 | 0 | 0
  Rel Fever | 15 | 31 | 27
  G3 Rel Fever | 0 | 0 | 0
  MA Fever | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: as for outcome 18
Time Frame: During the 4-day (Days 0-3) post-vaccination period following Dose 2.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 182 | 184 | 179
Participants
  Any Drowsiness | 97 | 132 | 109
  ≥ G 2 Drowsiness | 31 | 43 | 39
  G 3 Drowsiness | 8 | 7 | 4
  Rel Drowsiness | 94 | 126 | 108
  G3 Rel Drowsiness | 7 | 7 | 3
  MA Drowsiness | 0 | 0 | 0
  Any Irritability / Fussiness | 128 | 147 | 136
  ≥ G 2 Irritability / Fussiness | 53 | 70 | 61
  G 3 Irritability / Fussiness | 6 | 14 | 11
  Rel Irritability / Fussiness | 125 | 143 | 133
  G3 Rel Irritability / Fussiness | 6 | 13 | 11
  MA Irritability / Fussiness | 0 | 0 | 2
  Any Loss of appetite | 56 | 55 | 56
  ≥ G 2 Loss of appetite | 17 | 15 | 15
  G 3 Loss of appetite | 1 | 1 | 2
  Rel Loss of appetite | 52 | 51 | 55
  G3 Rel Loss of appetite | 1 | 1 | 2
  MA Loss of appetite | 0 | 0 | 1
  Any Fever | 47 | 36 | 35
  ≥ G 2 Fever | 2 | 3 | 2
  G 3 Fever | 0 | 0 | 0
  Rel Fever | 37 | 32 | 33
  G3 Rel Fever | 0 | 0 | 0
  MA Fever | 0 | 0 | 0

20. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: The solicited general symptoms assessed were Drowsiness, Irritability/Fussiness, Loss Of Appetite and Fever (defined as temperature ≥ 38.0°C). Any = any reports of the specific symptom irrespective of intensity grade; Grade 2 (G2) Drowsiness = Drowsiness that interfered with normal activity; Grade 2 Irritability/Fussiness = Moderate: Cried more than usual/interfered with normal activity; Grade 2 Loss of appetite = Ate less than usual/interfered with normal activity; Grade 2 Feve:r > 39.0 °C; Grade 3 (G3) Drowsiness/Irritability/Fussiness = symptom that prevented normal activity; Grade 3 Loss of appetite = Did not eat at all; Grade 3 Fever: > 40.0 °C; Related (Rel) = Symptom which was assessed by the investigator as related to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following Dose 3.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 172 | 175 | 170
Participants
  Any Drowsiness | 85 | 108 | 88
  ≥ G 2 Drowsiness | 23 | 37 | 25
  G 3 Drowsiness | 3 | 5 | 9
  Rel Drowsiness | 81 | 105 | 86
  G3 Rel Drowsiness | 3 | 5 | 9
  MA Drowsiness | 0 | 2 | 1
  Any Irritability / Fussiness | 126 | 135 | 122
  ≥ G 2 Irritability / Fussiness | 46 | 58 | 58
  G 3 Irritability / Fussiness | 6 | 15 | 11
  Rel Irritability / Fussiness | 121 | 129 | 120
  G3 Rel Irritability / Fussiness | 6 | 13 | 11
  MA Irritability / Fussiness | 0 | 3 | 1
  Any Loss of appetite | 45 | 58 | 53
  ≥ G 2 Loss of appetite | 11 | 13 | 15
  G 3 Loss of appetite | 1 | 2 | 2
  Rel Loss of appetite | 44 | 56 | 52
  G3 Rel Loss of appetite | 1 | 2 | 2
  MA Loss of appetite | 0 | 1 | 0
  Any Fever | 40 | 45 | 37
  ≥ G 2 Fever | 4 | 11 | 7
  G 3 Fever | 0 | 2 | 0
  Rel Fever | 35 | 39 | 35
  G3 Rel Fever | 0 | 2 | 0
  MA Fever | 1 | 2 | 1

21. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: as for outcome 18
Time Frame: During the 4-day (Days 0-3) post-vaccination period following any dose.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 187 | 189 | 188
Participants
  Any Drowsiness | 147 | 172 | 168
  ≥ G 2 Drowsiness | 67 | 88 | 81
  G 3 Drowsiness | 11 | 19 | 22
  Rel Drowsiness | 144 | 169 | 166
  G3 Rel Drowsiness | 11 | 18 | 21
  MA Drowsiness | 1 | 2 | 1
  Any Irritability / Fussiness | 164 | 182 | 177
  ≥ G 2 Irritability / Fussiness | 96 | 128 | 120
  G 3 Irritability / Fussiness | 18 | 35 | 30
  Rel Irritability / Fussiness | 161 | 180 | 175
  G3 Rel Irritability / Fussiness | 18 | 34 | 30
  MA Irritability / Fussiness | 1 | 3 | 3
  Any Loss of appetite | 95 | 111 | 117
  ≥ G 2 Loss of appetite | 28 | 32 | 39
  G 3 Loss of appetite | 2 | 3 | 6
  Rel Loss of appetite | 91 | 108 | 116
  G3 Rel Loss of appetite | 2 | 3 | 6
  MA Loss of appetite | 0 | 1 | 1
  Any Fever | 72 | 78 | 72
  ≥ G 2 Fever | 6 | 14 | 10
  G 3 Fever | 0 | 2 | 0
  Rel Fever | 61 | 74 | 69
  G3 Rel Fever | 0 | 2 | 0
  MA Fever | 1 | 2 | 1

22. Secondary Outcome: Number of Subjects With Specific Adverse Events (AEs).
Description: Occurrence of specific adverse events, i.e., new onset chronic diseases (e.g. autoimmune disorders, asthma, type I diabetes and allergies)
Time Frame: From Month 0 up to 6 months post primary-vaccination (Month 10)
Population: The analysis was done on the Primary Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 195 | 194 | 196
Participants | 7 | 11 | 10

23. Secondary Outcome: Number of Subjects With Unsolicited AEs.
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Days 0-30) post-primary vaccination period.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 195 | 194 | 196
Participants | 113 | 108 | 96

24. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs were defined as medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Month 0 up to 6 months post-primary vaccination (Month 10)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 195 | 194 | 196
Participants | 7 | 1 | 7

25. Secondary Outcome: Number of Seroprotected Subjects Against Anti-T.
Description: A seroprotected subject was defined a subject with antibody concentrations ≥ 0.1 IU/mL.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)] and at Visit 6 (At Month 14-17 one month after the booster dose (Dose 4)]
Population: The analysis was done on the Booster ATP cohort for immunogenicity, which included all subjects who complied with the protocol and study procedures up to the post-dose 4 blood sample and had immunogenicity results for the post-dose 4 blood sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 136 | 126
Participants
  Anti-T at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-T at Visit 5 | 118 | 123 | 107
  Anti-T at Visit 6 | 138 | 136 | 125

26. Secondary Outcome: Number of Seroprotected Subjects Against Anti-D.
Description: A seroprotected subject was defined a subject with antibody concentrations ≥ 0.1 IU/mL.
Time Frame: as for outcome 25
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 136 | 126
Participants
  Anti-D at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-D at Visit 5 | 128 | 123 | 115
  Anti-D at Visit 6 | 138 | 136 | 126

27. Secondary Outcome: Antibody Concentrations for Anti-T.
Description: Concentrations were expressed as GMCs for the seropositivity cut-off of 0.1 IU/mL.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)] and at Visit 6 [At Month 14-17 one month after the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 136 | 126
IU/mL
  Anti-T at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-T at Visit 5 | 0.327 [0.281 to 0.380] | 0.402 [0.340 to 0.474] | 0.340 [0.281 to 0.410]
  Anti-T at Visit 6 | 9.212 [7.863 to 10.793] | 8.870 [7.668 to 10.261] | 6.880 [5.905 to 8.015]

28. Secondary Outcome: Antibody Concentrations for Anti-D.
Description: Concentrations were expressed as GMCs for the seropositivity cut-off of 0.1 IU/mL.
Time Frame: as for outcome 27
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 136 | 126
IU/mL
  Anti-D at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-D at Visit 5 | 0.701 [0.597 to 0.825] | 0.622 [0.514 to 0.753] | 0.764 [0.629 to 0.928]
  Anti-D at Visit 6 | 8.334 [7.479 to 9.286] | 7.886 [6.972 to 8.92] | 8.537 [7.524 to 9.687]

29. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN.
Description: as for outcome 2
Time Frame: At Visit 5 [Month 13-16 before the booster dose (Dose 4)] and at Visit 6 [Month 14-17 one month after the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 136 | 126
Participants
  Anti-PT at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-PT at Visit 5 | 107 | 114 | 63
  Anti-FHA at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-FHA at Visit 5 | 130 | 130 | 113
  Anti-PRN at Visit 5: number analyzed (Participants) | 131 | 132 | 120
  Anti-PRN at Visit 5 | 110 | 104 | 91
  Anti-PT at Visit 6 | 138 | 136 | 126
  Anti-FHA at Visit 6 | 138 | 136 | 126
  Anti-PRN at Visit 6: number analyzed (Participants) | 137 | 136 | 125
  Anti-PRN at Visit 6 | 136 | 136 | 124

30. Secondary Outcome: Antibody Concentrations for Anti-PT, Anti-FHA and Anti-PRN.
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the following cut-offs:2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA, and 2.187 IU/mL for anti-PRN.
Time Frame: as for outcome 29
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 136 | 126
IU/mL
  Anti-PT Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-PT Visit 5 | 5.3 [4.6 to 6.2] | 6.5 [5.6 to 7.7] | 3.1 [2.6 to 3.7]
  Anti-FHA Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-FHA Visit 5 | 17.1 [14.7 to 19.9] | 21.8 [18.3 to 26.1] | 8.1 [6.6 to 9.9]
  Anti-PRN Visit 5: number analyzed (Participants) | 131 | 132 | 120
  Anti-PRN Visit 5 | 6.8 [5.5 to 8.3] | 5.5 [4.5 to 6.6] | 6.0 [4.8 to 7.5]
  Anti-PT Visit 6 | 71.4 [62.6 to 81.5] | 87.6 [76.6 to 100.2] | 55.5 [47.4 to 65.1]
  Anti-FHA Visit 6 | 186.9 [165.1 to 211.5] | 250.4 [220.4 to 284.6] | 101.0 [86.2 to 118.3]
  Anti-PRN Visit 6: number analyzed (Participants) | 137 | 136 | 125
  Anti-PRN Visit 6 | 208.0 [172.3 to 251.1] | 215.6 [176.1 to 263.8] | 130.5 [105.9 to 160.9]

31. Secondary Outcome: Number of Subjects With a Booster Response for Anti-PT, Anti-FHA and Anti-PRN.
Description: Booster response to PT, FHA and PRN antigens was defined as:
  * For subjects with pre-vaccination antibody concentration below the assay cut off, post-vaccination antibody concentration equal or above 4 times the assay cut-off.
  * For subjects with pre-vaccination antibody concentration between the assay cut off and below 4 times the assay cut-off, post-vaccination antibody concentration equal or above 4 times the pre-vaccination antibody concentration.
  * For subjects with pre-vaccination antibody concentration equal or above 4 times the assay cut-off, post-vaccination antibody concentration of at least two times the pre-vaccination antibody concentration.
  The assay cut off is 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA, and 2.187 IU/mL for anti-PRN.
Time Frame: At Visit 6 [At Month 14-17 one month after the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 131 | 130 | 116
Participants
  Anti-PT | 126 | 121 | 111
  Anti-FHA | 130 | 127 | 114
  Anti-PRN: number analyzed (Participants) | 130 | 130 | 115
  Anti-PRN | 128 | 128 | 112

32. Secondary Outcome: Number of Seroprotected Subjects Against Anti-PRP.
Description: A seroprotected subject was defined as a subject with anti-PRP concentrations ≥ 0.15 µg/mL.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)] and at Visit 6 [At Month 14-17 one month after the booster dose (Dose4)]
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 139 | 131
Participants
  Anti-PRP at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-PRP at Visit 5 | 91 | 122 | 94
  Anti-PRP at Visit 6 | 138 | 139 | 129

33. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 1 µg/mL.
Description: The cut-off for this assay was an anti-PRP concentration ≥ 1 µg/mL.
Time Frame: as for outcome 32
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 139 | 131
Participants
  Anti-PRP at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-PRP at Visit 5 | 23 | 71 | 47
  Anti-PRP at Visit 6 | 136 | 138 | 128

34. Secondary Outcome: Antibody Concentrations for Anti-PRP.
Description: Antibody concentrations were expressed as GMCs for the seroprotection cut-off of 1 µg/mL.
Time Frame: as for outcome 27
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 138 | 139 | 131
µg/mL
  Anti-PRP at Visit 5: number analyzed (Participants) | 131 | 132 | 121
  Anti-PRP at Visit 5 | 0.301 [0.242 to 0.373] | 0.987 [0.775 to 1.256] | 0.614 [0.458 to 0.822]
  Anti-PRP at Visit 6 | 39.365 [31.520 to 49.164] | 51.140 [41.954 to 62.339] | 27.318 [21.140 to 35.302]

35. Secondary Outcome: Number of Seroprotected Subjects Against Anti-polio Types 1, 2 and 3.
Description: A seroprotected subject was defined as a subject with anti-polio types 1, 2 and 3 titres ≥ 8 dilution.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 128 | 129 | 117
Participants
  Anti-polio 1: number analyzed (Participants) | 128 | 128 | 116
  Anti-polio 1 | 124 | 121 | 100
  Anti-polio 2: number analyzed (Participants) | 128 | 128 | 117
  Anti-polio 2 | 119 | 122 | 109
  Anti-polio 3: number analyzed (Participants) | 127 | 129 | 117
  Anti-polio 3 | 123 | 126 | 80

36. Secondary Outcome: Antibody Titres for Anti-polio Types 1, 2 and 3.
Description: Titres were expressed as geometric mean titres (GMTs) for the cut-off of 8 dilution.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: titres
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 128 | 129 | 117
titres
  Anti-polio 1: number analyzed (Participants) | 128 | 128 | 116
  Anti-polio 1 | 99.5 [79.4 to 124.8] | 107.4 [83.7 to 137.9] | 42.2 [32.6 to 54.6]
  Anti-polio 2: number analyzed (Participants) | 128 | 128 | 117
  Anti-polio 2 | 94.9 [73.2 to 123.1] | 111.9 [88.0 to 142.4] | 51.2 [40.8 to 64.3]
  Anti-polio 3: number analyzed (Participants) | 127 | 129 | 117
  Anti-polio 3 | 122.1 [95.1 to 156.9] | 160.4 [125.8 to 204.6] | 28.4 [20.6 to 39.1]

37. Secondary Outcome: Number of Seroprotected Subjects Against Anti-HBs.
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 133 | 131 | 121
Participants | 131 | 128 | 105

38. Secondary Outcome: Antibody Concentrations for Anti-HBs.
Description: Antibody concentrations were expressed as GMCs for the seroprotection cut-off of 10 mIU/mL.
Time Frame: At Visit 5 [At Month 13-16 before the booster dose (Dose 4)]
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 133 | 131 | 121
mIU/mL | 328.7 [261.5 to 413.2] | 235.8 [188.2 to 295.5] | 149.4 [100.5 to 222.3]

39. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: as for outcome 17
Time Frame: During the 4-day (Days 0-3) post-booster vaccination.
Population: The analysis was done on the Booster Total Vaccinated cohort, which included all subjects with documented administration of the booster vaccine and with the symptoms sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 154 | 151 | 150
Participants
  Any Pain, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  Any Pain, ActHIB/Hiberix | 61 | 64 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  ≥ G 2 Pain, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  ≥ G 2 Pain, ActHIB/Hiberix | 11 | 15 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  G 3 Pain, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  G 3 Pain, ActHIB/Hiberix | 1 | 2 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  MA Pain, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  MA Pain, ActHIB/Hiberix | 0 | 0 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  Any Pain, Infanrix/Pentacel | 62 | 74 | 59
  ≥ G2 Pain, Infanrix/Pentacel | 12 | 19 | 16
  G3 Pain, Infanrix/Pentacel | 2 | 3 | 2
  MA Pain, Infanrix/Pentacel | 1 | 0 | 0
  Any Red, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  Any Red, ActHIB/Hiberix | 42 | 49 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  ≥ G 2 Red, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  ≥ G 2 Red, ActHIB/Hiberix | 7 | 4 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  G 3 Red, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  G 3 Red, ActHIB/Hiberix | 0 | 2 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  MA Red, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  MA Red, ActHIB/Hiberix | 0 | 0 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  Any Red, Infanrix/Pentacel | 49 | 60 | 47
  ≥ G2 Red, Infanrix/Pentacel | 17 | 14 | 13
  G3 Red, Infanrix/Pentacel | 8 | 4 | 2
  MA Red, Infanrix/Pentacel | 2 | 0 | 0
  Any Swe, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  Any Swe, ActHIB/Hiberix | 29 | 29 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  ≥ G 2 Swe, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  ≥ G 2 Swe, ActHIB/Hiberix | 7 | 6 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  G 3 Swe, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  G 3 Swe, ActHIB/Hiberix | 0 | 2 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  MA Swe, ActHIB/Hiberix: number analyzed (Participants) | 153 | 151 | 150
  MA Swe, ActHIB/Hiberix | 0 | 0 | NA — Subjects in Pentacel Group did not receive the ActHIB or Hiberix vaccines.
  Any Swe, Infanrix/Pentacel | 42 | 44 | 35
  ≥ G2 Swe, Infanrix/Pentacel | 13 | 17 | 14
  G3 Swe, Infanrix/Pentacel | 5 | 7 | 4
  MA Swe, Infanrix/Pentacel | 2 | 0 | 0

40. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: The solicited general symptoms assessed were Drowsiness, Irritability/Fussiness, Loss Of Appetite and Fever (defined as temperature ≥ 38.0°C). Any = any reports of the specific symptom irrespective of intensity grade; Grade 2 (G2) Drowsiness = Drowsiness that interfered with normal activity; Grade 2 Irritability/Fussiness = Moderate: Cried more than usual/interfered with normal activity; Grade 2 Loss of appetite = Ate less than usual/interfered with normal activity; Grade 2 Fever: > 39.0 °C and ≤ 40.0 °C; Grade 3 (G3) Drowsiness/Irritability/Fussiness = symptom that prevented normal activity; Grade 3 Loss of appetite = Did not eat at all; Grade 3 Fever: > 40.0 °C; Related (Rel) = Symptom which was assessed by the investigator as related to vaccination.
Time Frame: During the 4-day (Days 0-3) post-booster vaccination.
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 153 | 150 | 151
Participants
  Any Drowsiness | 59 | 67 | 65
  ≥ G 2 Drowsiness | 18 | 20 | 17
  G 3 Drowsiness | 1 | 3 | 2
  Rel Drowsiness | 55 | 65 | 61
  G3 Rel Drowsiness | 1 | 3 | 2
  MA Drowsiness | 0 | 0 | 0
  Any Irritability / Fussiness | 86 | 94 | 76
  ≥ G 2 Irritability / Fussiness | 26 | 35 | 23
  G 3 Irritability / Fussiness | 3 | 4 | 4
  Rel Irritability / Fussiness | 85 | 92 | 68
  G3 Rel Irritability / Fussiness | 3 | 4 | 4
  MA Irritability / Fussiness | 0 | 0 | 1
  Any Loss of appetite | 47 | 47 | 46
  ≥ G 2 Loss of appetite | 8 | 9 | 11
  G 3 Loss of appetite | 1 | 2 | 2
  Rel Loss of appetite | 44 | 44 | 41
  G3 Rel Loss of appetite | 1 | 2 | 2
  MA Loss of appetite | 0 | 0 | 0
  Any Fever | 4 | 10 | 11
  ≥ G 2 Fever | 1 | 1 | 1
  G 3 Fever | 0 | 0 | 0
  Rel Fever | 2 | 10 | 9
  G3 Rel Fever | 0 | 0 | 0
  MA Fever | 0 | 2 | 1

41. Secondary Outcome: Number of Subjects With Specific AEs.
Description: as for outcome 22
Time Frame: During the 31-day (Days 0-30) post-booster vaccination.
Population: The analysis was done on the Booster Total Vaccinated cohort, which included all subjects with documented administration of the booster vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 167 | 158 | 161
Participants | 4 | 1 | 1

42. Secondary Outcome: Number of Subjects With Unsolicited AEs.
Description: as for outcome 23
Time Frame: During the 31-day (Days 0-30) post-booster vaccination.
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 167 | 158 | 161
Participants | 37 | 35 | 41

43. Secondary Outcome: Number of Subjects With SAEs.
Description: as for outcome 24
Time Frame: During the 31-day (Days 0-30) post-booster vaccination.
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
Number analyzed (Participants) | 167 | 158 | 161
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Day 0-Day 3) follow-up period after each dose. Unsolicited AEs: during the 31-day (Day 0-Day 30) follow-up period after each dose. SAEs: during the entire study period (from Month 0 to Month 17).
Arm/Group | Infanrix Hexa Group | Pediarix Group | Pentacel Group
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/194 | 0/196
Serious Adverse Events (participants affected / at risk) | 8/195 | 1/194 | 8/196
Other Adverse Events (participants affected / at risk) | 188/195 | 190/194 | 187/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix Hexa Group (N=195) | Pediarix Group (N=194) | Pentacel Group (N=196)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix Hexa Group (N=195) | Pediarix Group (N=194) | Pentacel Group (N=196)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Asymmetric gluteal fold (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Candida nappy rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 3 (3) | 1 (1)
Conjunctivitis (Infections and infestations) | 10 (10) | 9 (10) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 8 (8) | 7 (7)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Crying (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Dacryostenosis acquired (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 112 (201) | 126 (236) | 127 (235)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8) | 7 (7)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 10 (11)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 7 (7) | 13 (14)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 4 (4)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 8 (8) | 1 (1)
Genital labial adhesions (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Herpangina (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 2 (2) | 5 (5)
Injection site erythema (General disorders) | 112 (228) | 129 (299) | 116 (248)
Injection site induration (General disorders) | 3 (4) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 141 (322) | 162 (423) | 152 (361)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 2 (3)
Injection site scab (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 92 (166) | 103 (201) | 90 (180)
Injection site warmth (General disorders) | 0 (0) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 167 (461) | 183 (544) | 180 (488)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 2 (2) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 2 (2)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 10 (10) | 11 (13) | 12 (12)
Otitis media acute (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Penile adhesion (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 0 (0)
Penile erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Plagiocephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Positional plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 82 (133) | 85 (136) | 82 (130)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8) | 6 (6)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5) | 5 (6)
Roseola (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Screaming (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 152 (355) | 173 (450) | 173 (411)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 8 (10) | 10 (11) | 11 (12)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 32 (35) | 26 (31) | 32 (35)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Vaccination site bruising (General disorders) | 0 (0) | 2 (3) | 1 (1)
Vaccination site erythema (General disorders) | 2 (2) | 5 (5) | 3 (3)
Vaccination site induration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 2 (2) | 1 (1) | 3 (3)
Vaccination site swelling (General disorders) | 3 (3) | 1 (1) | 2 (2)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 4 (4) | 3 (3) | 8 (8)
Viral rash (Infections and infestations) | 3 (3) | 0 (0) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 13 (13) | 10 (11) | 12 (12)
Vomiting projectile (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.